CLINICAL TRIAL: NCT05837806
Title: A Single-arm, Open Clinical Trial of Efficacy and Safety of Tislelizumab in Combination With Disitamab-vedotin as Neoadjuvant Therapy for HER2-positive High-risk Upper Tract Urothelial Carcinoma (UTUC)
Brief Title: Efficacy and Safety of Tislelizumab in Combination With Disitamab-vedotin as Neoadjuvant Therapy for HER2-positive High-risk Upper Tract Urothelial Carcinoma (UTUC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRUCE-UTUC01
Record Dates: First submitted 2023-04-14; First posted 2023-05-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-06

CONDITIONS: Neoadjuvant Immunotherapy
Keywords: neoadjuvant therapy; UTUC; immunotherapy; upper tract urothelial carcinoma; PD-1; ADC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tislelizumab+disitamab-vedotin (Experimental)
  Interventions: Drug: tislelizumab+disitamab-vedotin

INTERVENTIONS:
Drug: tislelizumab+disitamab-vedotin — Patients enrolled will receive 3 cycles of tislelizumab 200 mg in combination with disitamab-vedotin (RC48) 2.0mg/kg intravenously.

SUMMARY:
Neoadjuvant chemotherapy treatment can be used for specific UTUC patients, especially for highly staged and/or grade tumors, such as kidneys with potentially decreased renal function after RNU. Neoadjuvant therapy is a series of treatments administered preoperatively for UTUC, mainly chemotherapy, and in recent years, novel therapies of immunotherapy have emerged. Since conventional cisplatin neoadjuvant regimens also require high preoperative renal function, neoadjuvant therapy regimens such as immunotherapy provide more effective and feasible treatments for patients who are intolerant to current cisplatin chemotherapy regimens. The aim of this study was to explore the efficacy and safety of the combination of disitamab vedotin, a human epidermal growth factor receptor-2 (HER-2) targeted ADC, and tislelizumab, a humanised PD-1 ICIs, as neoadjuvant treatment for non-metastatic, high-risk, HER-2 expressing UTUC. In our study, patients enrolled will receive neoadjuvant tislelizumab plus disitamab-vedotin therapy followed by radical nephroureterectomy (RNU), distal ureterectomy (DU) or ureteroscopic ablation (UA) .

ELIGIBILITY:
Inclusion Criteria:

1. Radiographically(CT, MRI or PET-CT, etc.) and histologically confirmed diagnosis of localized HER-2 expressing upper urothelial carcinoma( (cT1-4N0-2M0, HER-2 immunohistochemistry (IHC) ≥ 1+); high risk disease (according to EAU Guidelines for UTUC); planning to receive radical nephroureterectomy (RNU), distal ureterectomy (DU) or ureteroscopic ablation (UA).
2. Male or female aged 18 years and above;
3. Expected survival time greater than 12 weeks;
4. An ECOG status score of 0-2;
5. Agree to provide specimens of blood, urine, and tissue examination (for detection of MRD, PD-L1 expression, HER2 expression, tumor mutation load, immunohistochemistry, DNA and RNA detection, etc.);
6. The level of organ function must meet the following requirements:

   * hematological indicators: absolute neutrophil count ≥ 1.5 × 10^9/L, platelet count ≥ 80 × 10^9/L, hemoglobin ≥ 6.0 g/dL (can be maintained by symptomatic treatment)
   * hepatic function: total bilirubin ≤ 1.5 times the upper limit of normal, and glutathione and glutamic oxalacetic transaminase ≤ 2.5 times the upper limit of normal;
   * renal function: GFR ≥ 15 ml/min;
   * Subjects voluntarily joined the study, signed an informed consent form, were compliant, and cooperated with the follow-up.

Exclusion Criteria:

1. Live attenuated vaccines, other than COVID-19 vaccine, received within 4 weeks prior to treatment or scheduled to be received during the study period
2. Active, known or suspected autoimmune disease;
3. Known history of primary immunodeficiency;
4. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
5. Female patients who are pregnant or breastfeeding
6. Untreated acute or chronic active hepatitis B or C infection. Patients who are receiving antiviral therapy with monitoring of viral copy number and are eligible for enrollment as determined by the physician on an individual patient basis;
7. Previous use of immunosuppressive drugs, excluding nasal spray and inhaled corticosteroids or physiologic doses of systemic steroids (i.e., no more than 10 mg/day prednisolone or equivalent pharmacologic physiologic doses of other corticosteroids), within 4 weeks prior to initiation of therapy
8. Known or suspected allergy history to tislelizumab and disitamab vedotin.
9. With a clear history of active tuberculosis.
10. Prior PD-1/PD-L1/CTLA-4 antibody or other immunotherapy;
11. Those who are participating in other clinical studies
12. Men of reproductive potential or women with the potential to become pregnant who are not using reliable contraception
13. Uncontrolled co-morbidities, including but not limited to

    * HIV-infected individuals (HIV-positive);
    * Severe infections that are active or poorly controlled clinically (including patients in the period of neocoronavirus infection)
    * Evidence of the presence of severe or uncontrolled systemic disease (e.g., severe psychiatric, neurological disease, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, hepatic or renal disease, uncontrolled hypertension [i.e., defined as greater than or equal to CTCAE grade 2 hypertension despite medication]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) | 3 months
  no residual lesions were found in the imaging examination, negative urine cytology and pathological examination showed no tumor was detected in the specimen from radical nephroureterectomy (RNU), distal ureterectomy (DU) or ureteroscopic ablation (UA).

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Hu, MD,PhD, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- The Second Hospital of Tianjin Medical University, Tianjin, China